CLINICAL TRIAL: NCT06394856
Title: Comparison of Outcomes of Rotator Cuff Repair With a Modified Versus Classic Double-Row Suture -Bridge Techniques
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Hossam Eldin Mohamed Ahmed ElAzab, assistant professor orthopedic department, Sohag University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Soh-Med-23-04-01
Record Dates: First submitted 2024-04-21; First posted 2024-05-01 (Actual); Last update posted 2024-06-13 (Actual); Status verified 2024-06

CONDITIONS: Rotator Cuff Tears
MeSH Terms: conditions — Rotator Cuff Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- knotless group (Active Comparator): rotator cuff repair with a modified knotless anchors
  Interventions: Procedure: Rotator Cuff Repair With a Modified Versus Classic Double-Row Suture -Bridge Techniques
- knot-tying group (Active Comparator): rotator cuff repair with classic knot-tying double-row suture bridge technique by classic anchors
  Interventions: Procedure: Rotator Cuff Repair With a Modified Versus Classic Double-Row Suture -Bridge Techniques

INTERVENTIONS:
Procedure: Rotator Cuff Repair With a Modified Versus Classic Double-Row Suture -Bridge Techniques — rotator cuff tears with modified versus classic double row suture bridge

SUMMARY:
rotator cuff tears are one of the most common shoulder issues , affecting 20.7% of the general population .

DETAILED DESCRIPTION:
accompanied by shoulder pain and dysfunction

ELIGIBILITY:
Inclusion Criteria:

* full-thickness supraspinatus
* degenerative tears
* age range 40 :65

Exclusion Criteria:

* subscapularis tear
* small and massive tears
* traumatic tears
* partial -thickness tear
* revisioin surgery
* glenohumeral arthretic changes and shoulder instability

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2021-07-01 (Actual)

PRIMARY OUTCOMES:
retear rate | 3 years
  retear rate

SECONDARY OUTCOMES:
time | 3 years
  duration of operation

CONTACTS AND LOCATIONS:
Overall Officials: Hossam M azab, MD, Study Chair — Sohag University
Locations (1):
- university Hospital, Sohag, Egypt